CLINICAL TRIAL: NCT04181931
Title: Neoadjuvant Transartery Chemoembolization Plus Artery Infusion Chemotherapy With Surgery Versus Surgery Alone for Hepatocellular Carcinoma Patients With Portal Vein Tumor Thrombus: a Randomized Clinical Trial
Brief Title: Neo-TACE-HAIC for PVTT-HCC
Acronym: NeoconceptC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-170
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neo-TACE-HAIC with surgery (Experimental): neoadjuvant TACE-HAIC with surgery for HCC patients with PVTT
  Interventions: Procedure: neo-TACE-HAIC+Surgery
- surgery alone (Active Comparator): surgery alone for HCC patients with PVTT
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Procedure: neo-TACE-HAIC+Surgery — transartery chemoembolization with lipiodol and EADM, FOLFOX (Oxa 85mg/m2 2h+CF 400mg/m2 2h+5FU 400mg/m2 10min+5FU 1200mg/m2 23h)-based artery infusion chemotherapy, followed by hepatic resection
  Arms: neo-TACE-HAIC with surgery
Procedure: Surgery alone — hepatic resection remove the liver tumor and portal vein tumor thrombus
  Arms: surgery alone

SUMMARY:
Hepatocellular carcinoma (HCC) patients is a common disease in the East Asia. During the disease course, 20%-50% patients suffered portal vein tumor thrombus (PVTT), which is characterized with poor outcome and low response for treatments. Although BCLC (Barcelona clinical liver cancer) system recommend to palliative targeted treatment, the East Asian countries recommend to resection or transartery chemoembolization (TACE).

Recently, FOLFOX (Oxaliplatin and 5-fluorouracil) based hepatic artery infusion chemotherapy (HAIC) exhibited high response rate for advanced HCC.

Pilot study showed TACE combined HAIC (TACE-HAIC) had better tumor response, with low progression disease rate.

Whether TACE-HAIC would improve survival for patients with PVTT is need to further to study. A randomized clinical trial compared neo-TACE-HAIC with surgery versus surgery alone is aimed to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;
* Patients with resectable primary hepatocellular carcinoma and portal vein tumor thrombus, which was not located in main portal vein;
* Child-Pugh A or B (7 score) liver function;
* With more than 3 months expected survival;
* The volume of residual liver more than 30%

Exclusion Criteria:

* Patients with primary hepatocellular carcinoma and major portal vein tumor thrombus
* With extrahepatic metastasis or unresectable HCC
* Pregnant woman or sucking period;
* With other malignant cancer;
* Received chemotherapy, target therapy or immunosuppressive drugs therapy before this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | 36 months
  PFS was calculated from the date of starting treatment to the date of progression, of disease or death.

SECONDARY OUTCOMES:
Overall survival, OS | 60 months
  OS was calculated from the date of starting treatment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No